CLINICAL TRIAL: NCT05735262
Title: Personalized Brain Functional Sectors (pBFS) Guided Precision Neuromodulation Treatment for Autism Spectrum Disorder (ASD): a Single-center, Sham-controlled, Double-blinded, Randomized Clinical Trial Study
Brief Title: pBFS Guided Precision Neuromodulation Treatment for ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changping Laboratory (Other)
Collaborators: China Rehabilitation Research Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPASD2023BA100
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-02

CONDITIONS: Autism Spectrum Disorder
Keywords: TMS, fMRI, ASD, personalized
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DLPFC group (Experimental): Active iTBS will be delivered to the left DLPFC.
  Interventions: Device: active iTBS
- DMPFC group (Experimental): Active iTBS will be delivered to the left DMPFC.
  Interventions: Device: active iTBS
- Sham to DLPFC group (Sham Comparator): Sham iTBS will be delivered to left DLPFC.
  Interventions: Device: sham iTBS
- Sham to DMPFC group (Sham Comparator): Sham iTBS will be delivered to left DMPFC.
  Interventions: Device: sham iTBS

INTERVENTIONS:
Device: active iTBS — Each participant will receive 1800 pulse active iTBS (100% RMT) in each session, 3 sessions per day, 5 days per week for 8 weeks.
  Arms: DLPFC group; DMPFC group
Device: sham iTBS — Each participant will receive 1800 pulse sham iTBS (100% RMT) in each session, 3 sessions per day, 5 days per week for 8 weeks.
  Arms: Sham to DLPFC group; Sham to DMPFC group

SUMMARY:
This study aims to evaluate the neuromodulation (i.e., iTBS) effectiveness for treating autism spectrum disorder (ASD) by targeting at the pBFS-guided executive function brain network or social brain network.

DETAILED DESCRIPTION:
Autism spectrum disorder is characterized by executive function deficiency and social interaction difficulty. Using the developed technique, personalized brain functional sectors (pBFS), we could precisely identify individualized brain function networks based on the resting-state functional MRI scan. A tailored dorsal lateral prefrontal cortex (DLPFC) region situated within the executive function network and a tailored dorsal medial prefrontal cortex (DMPFC) region situated within the social network will be selected as intervention targets.

The participants will be equally randomized to the following three groups, active iTBS to the left DLPFC, active iTBS to the left DMPFC, and sham iTBS to either the left DLPFC or left DMPFC at a ratio of 2:2:1:1. Each participant will receive 1800 pulse active or sham iTBS (100% RMT) in each session, 3 sessions daily, 5 days per week for 8 weeks, as well as background behavioral training between iTBS sessions.

ELIGIBILITY:
Inclusion Criteria:

* 6-30 years old
* Have the diagnosis of autism spectrum disorder
* ADOS-2 score is higher than the ASD cut-offs
* Capacity to follow the study procedures, including fMRI scan under sedation, assessment, and rehabilitation training
* Participant's parents or other legal guardians give informed consent

Exclusion Criteria:

* Current or history of psychotic disorders, such as schizophrenia, bipolar disorder
* Severe self-injury or suicidal behavior presented in the last 1 year
* Severe visual, auditory, or motor disability that interferes with any study procedure
* Current, history or family history of epilepsy
* Known severe physical diseases, such as congenital heart defects, traumatic brain injury
* Metal implantations, which are contradicted by MRI or TMS, such as artificial cardiac pacemakers, stents, cochlear implants
* Received TMS, tCS, FUS, or other neuromodulation treatment in the last 3 months
* Currently participating in other clinical trials

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
ADOS-2 SA change | Pre-treatment (baseline), immediately post-treatment
  The social affect (SA) dimension score change of autism diagnostic observation scale, 2nd edition (ADOS-2) from baseline

SECONDARY OUTCOMES:
ADOS-2 total score change | Pre-treatment (baseline), immediately post-treatment
  The total score change of autism diagnostic observation scale, 2nd edition (ADOS-2) from baseline
CBCL score change | Pre-treatment (baseline), immediately post-treatment
  Score change of the child behavior checklist (CBCL) from baseline

OTHER OUTCOMES:
SRS-2 score change | Pre-treatment (baseline), immediately post-treatment
  Sore change of the Social Responsiveness Scale, 2nd edition (SRS-2) from baseline
RBS-R score change | Pre-treatment (baseline), immediately post-treatment
  Score change of the Repetitive Behavior Scale-Revised (RBS-R) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory
Locations (1):
- China Rehabilitation Research Center, Beijing, China